CLINICAL TRIAL: NCT03482843
Title: Vitamin D Effect on Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Clinic Frankfurt (Other)
Collaborators: Institut für Kardiovaskuläre Physiologie, Vascular Research Center (Unknown)
Responsible Party: Principal Investigator, Juergen Konczalla, Prof. Dr., University Clinic Frankfurt
Other Study IDs: 142/15
Record Dates: First submitted 2018-03-18; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin D Deficiency: 25-Vitamin D level <25 ng/ml
- Sufficient Vitamin D Level: 25-Vitamin D Level >=25-70 ng/ml

SUMMARY:
Vitamin D has been promoted to vascular regeneration in non-cerebral arteries because of its anti-inflammatory properties. Cerebral vasospasm (CVS) as the most feared complication after subarachnoid hemorrhage (SAH), correlated with higher mortality and poor outcome, is the result of a multifactorial mechanism with inflammation as one of the main role players. The investigators therefore hypothesized that vitamin D attenuates cerebral vasospasm and increases the chance for favorable outcome after SAH.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) as a worldwide significant cause for morbidity and mortality, especially affecting young population, accounts for 4%-10% of all strokes. About 25% of SAH patients die and 50% left with significant disability, which according to the relative youth of the affected individuals means that this event is responsible for a quarter of all years of life lost as a result of stroke. Cerebral vasospasm, as the most feared complication after SAH leading mostly into ischemia, associated with delayed deterioration, continues to be both a difficult entity to treat and a leading cause of morbidity in patients. A high number of investigators focused on vasospasm research to develop effective therapy strategies to treat this entity, however, results of experimental studies and clinical trials about calcium channel blocker nicardipine and the endothelin-1 antagonist clazosentan as sources of hope in vasospasm treatment did not reveal an improvement in patient outcomes. Recently, there is a renewed interest in looking for other potentially targets for therapy.

Vitamin D, especially the aktive hormone 1,25-dihydroxycholecalciferol (1,25VitD3), has been suggested to limit inflammation, cancer, development of heart failure and myocardial infarction through the nuclear vitamin D receptor (VDR) by balancing the gene expression. Thus, vitamin D deficiency is linked to increased risk in many clinical settings including cardiovascular disease, stroke and critically ill patients. Furthermore, low vitamin D status has been associated with autoimmune disorders such as multiple sclerosis or neoplastic diseases, increased rates of infections and increased mortality. In case of ischemic stroke, a higher rate of vitamin D insufficiency has been suggested in patients associated with poorer outcomes. Nevertheless, these observations still remain controversial.

However, current data attracted considerable attention in neurovascular research to study the effects of this hormone on SAH. Recently, a few experimental and clinical studies have already worked on this topic. A rat model of SAH confirmed that vitamin D pretreatment attenuates cerebral artery remodeling and vasospasm as well as blood-brain barrier (BBB) disruption mainly through endogenous upregulation of osteopontin. Clinical data proved the fact that there is an increased incidence of hypovitaminosis D among patients requiring treatment for cerebral aneurysms and a high prevalence of vitamin D insufficiency among SAH patients. Contrary to expectations, an association between vitamin D deficiency and outcomes in SAH patients could not be detected. However, in view of recent limited research data on this topic a final statement could not yet be made. Therefore, the investigators aimed to determine the effect of vitamin D on vasospasm discussing mechanistic evaluations of inflammation in SAH based on a translational study design including patient data to underline our experimental findings.

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients suffering from SAH over 18 years of age with consent form.

Exclusion Criteria:

* Admitted patients suffering from SAH younger than 18 years of age.
* SAH patients without consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All admitted SAH patients over 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical outcome at discharge | 2 to 4 weeks after SAH
  modified Rankin scale (for measuring the dependence in daily activity. Range 0 (no symptoms) to 6 (dead)

SECONDARY OUTCOMES:
clinical outcome 6 months after SAH | 6 months after SAH
  modified Rankin scale (for measuring the dependence in daily activity. Range 0 (no symptoms) to 6 (dead)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Konczalla, Prof., Principal Investigator — Goethe University Hospital
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Germany